CLINICAL TRIAL: NCT03557086
Title: A Randomized Controlled Trial of an Advanced Care Planning Video Decision Support Tool for Patients With End-Stage Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Nneka nnaoke Ufere, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018P001146
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Results first posted 2021-11-03 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: End Stage Liver Disease
MeSH Terms: conditions — End Stage Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Care Planning Video Decision Support Tool (Experimental): We designed a 3-minute advance care planning video to provide patients with advanced liver disease general understanding of the types of medical care patients may receive at the end of life (EOL) and a description of medical interventions such as hospitalizations, intensive care unit (ICU) admission, cardiopulmonary resuscitation (CPR), and intubation. The video begins by addressing the importance of the patient's personal goals and perspectives by asking the viewer to reflect on their concerns about getting sick and their overall goals for their EOL care. The physician narrator then introduces a framework for choices of medical care at the EOL including: 1) life-prolonging care; 2) limited medical care; and 3) comfort care followed by visual images illustrating each of these EOL care choices. All three sequences of video images accompanying the narration attempt to help the viewer imagine the experience and likely outcomes of receiving these medical interventions at the EOL.
  Interventions: Behavioral: Advance Care Planning Video Decision Support Tool
- Verbal Narrative Control (Active Comparator): Immediately after completing baseline assessments and randomization, patients assigned to the verbal narrative control arm will listen to the same description of the 3 goals of care used in the video arm read out by a research assistant
  Interventions: Other: Verbal Narrative

INTERVENTIONS:
Behavioral: Advance Care Planning Video Decision Support Tool — Advance care planning video intervention as previously described
  Arms: Advanced Care Planning Video Decision Support Tool
Other: Verbal Narrative — Verbal description of end of life care options
  Arms: Verbal Narrative Control

SUMMARY:
The goal of this pilot randomized trial is to assess the feasibility and preliminary efficacy of an advanced care planning (ACP) video decision support tool for improving patients' knowledge regarding their goals of care options and end of life (EOL) decision-making in patients with end-stage liver disease (ESLD).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age with an established diagnosis of end-stage liver disease
2. Patient must have either 1) primary hepatologist at the MGH Liver Center or an MGH-affiliated primary care physician, or 2) a previous inpatient admission at MGH
3. Deemed ineligible for liver transplantation as determined by the primary hepatologist
4. Ability to communicate in English and provide informed consent
5. A score ≥ 7 on the Short Portable Mental Status Questionnaire

Exclusion Criteria:

1. Severe hepatic encephalopathy which the primary hepatologist believes prohibits informed consent or participation in the study
2. Significant uncontrolled psychiatric disorders (psychotic disorder, bipolar disorder, major depression) or other co-morbid disease (dementia, cognitive impairment), which the primary hepatologist believes prohibits informed consent or participation in the study
3. Prior history of liver transplantation
4. Patient has been referred to or enrolled in hospice care
5. Patients who have been referred to palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ufere NN, Robinson B, Donlan J, Indriolo T, Bloom J, Scherrer A, Mason NM, Patel A, Lai JC, Chung RT, Volandes A, El-Jawahri A. Pilot Randomized Controlled Trial of an Advance Care Planning Video Decision Tool for Patients With Advanced Liver Disease. Clin Gastroenterol Hepatol. 2022 Oct;20(10):2287-2295.e3. doi: 10.1016/j.cgh.2021.10.027. Epub 2021 Oct 27. PMID 34718173

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Advanced Care Planning Video Decision Support Tool | Verbal Narrative Control
Started | 26 | 24
Completed | 26 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Advanced Care Planning Video Decision Support Tool | Verbal Narrative Control | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.5 [29 to 87] | 58.5 [40 to 66] | 60 [29 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 24 | 24 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  Some high school | 1 | 0 | 1
  High school graduate | 9 | 10 | 19
  Some college | 4 | 6 | 10
  College graduate | 9 | 5 | 14
  Postgraduate | 2 | 3 | 5
  Missing | 1 | 0 | 1
Marital Status [Count of Participants; unit: Participants]
  Married or with a partner | 17 | 14 | 31
  Widowed | 2 | 1 | 3
  Divorced | 4 | 6 | 10
  Single | 3 | 3 | 6
Model for End-Stage Liver Disease-Sodium (MELD-Na) Score [Median (Inter-Quartile Range); unit: units on a scale] — Model for End-Stage Liver Disease-Sodium (MELD-Na) Score is used to estimate relative liver disease severity. Scores range from 6 (minimum) to 40 (maximum) with higher scores associated with increasing severity of hepatic dysfunction and increased three-month mortality risk. The total score (and total score ranges) are reported.
  units on a scale | 16 [7 to 39] | 16.5 [7 to 35] | 16.5 [7 to 39]
Etiology of Liver Disease [Count of Participants; unit: Participants]
  Alcohol | 15 | 17 | 32
  NASH/Cryptogenic | 6 | 4 | 10
  Multifactorial/Other | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Eligible Participants Enrolled in the Study
Description: The proposed video intervention will be deemed feasible if at least 60% of eligible patients are enrolled in the study.
Time Frame: By 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Patients Approached for Enrollment Into the Study: We pre-specified the ACP video intervention as feasible if at least 60% of eligible patients enrolled in the study.
Arm/Group | Patients Approached for Enrollment Into the Study
Number analyzed (Participants) | 59
Participants | 50

2. Secondary Outcome: Changes in Knowledge Scores From Baseline to Post-intervention
Description: We will assess patients' knowledge of goals of care before and after the intervention using 5 true/false questions and 1 multiple choice question, each worth 1 point, for a summary score of 0 to 6 (higher score reflects greater knowledge). We have used this knowledge questionnaire in prior studies. Changes in knowledge scores from before and after the intervention will be compared between the intervention and control arms.
Time Frame: Baseline and post-intervention, by 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Advanced Care Planning Video Decision Support Tool | Verbal Narrative Control
Number analyzed (Participants) | 26 | 24
score on a scale | 5.7 (0.45) | 4.8 (0.76)

3. Secondary Outcome: Preferences for Life-prolonging Care, Preferences to Receive Cardiopulmonary Resuscitation (CPR), and Preferences to Receive Intubation
Description: Before and after the intervention, patients will report their post-intervention preferences for life-prolonging care: life-prolonging care, limited medical care, comfort care, or unsure. Before the intervention, patients will report their preferences to receive CPR as follows: "Yes, attempt CPR", "No, do not attempt CPR", or "Not sure." Before the intervention, patients will report their preferences to receive intubation as follows: "Yes, attempt intubation", "No, do not attempt intubation", or "Not sure."
  Post-intervention preferences for life-prolonging care (life-prolonging care, limited medical care, and comfort care), preferences to receive CPR, and preferences to receive intubation will be compared between the two groups.
Time Frame: By 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Care Planning Video Decision Support Tool | Verbal Narrative Control
Number analyzed (Participants) | 26 | 24
Participants
  Post-intervention preferences for life-prolonging care | 4 | 7
  Post-intervention preferences to receive CPR | 9 | 15
  Post-intervention preferences to receive intubation | 6 | 8

4. Secondary Outcome: Code Status Documentation
Description: Code status documentation in the electronic health record will be compared between the intervention and control arms.
Time Frame: By 12 months
Population: Data not collected due to lack of access to outside hospital electronic medical records to confirm code status documentation
Arm/Group | Advanced Care Planning Video Decision Support Tool | Verbal Narrative Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants Who Answered That They Felt "Very Comfortable" Seeing the Video in Response to First Question of Acceptability Questionnaire (Acceptability - Comfort)
Description: For the video intervention arm alone, we will administer 3-items assessing patients' comfort with watching the video, whether they find the video helpful in their understanding of the EOL care options, and whether they would recommend it to others. For the outcome of "comfort" we asked patients whether they felt comfortable watching the video by asking the question: "Did you feel comfortable seeing the video in order to help you answer the questions regarding medical care?". Response choices were on a Likert scale with answer choices as follows: 1) very comfortable; 2) somewhat comfortable; 3) not comfortable; 4) don't know. We report below the percentage of patients who answered "very comfortable".
Time Frame: By 12 months
Population: Patients randomized to the Advanced Care Planning Video Decision Support Tool intervention arm
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Care Planning Video Decision Support Tool
Number analyzed (Participants) | 26
Participants | 21

6. Secondary Outcome: Number of Participants Who Answered That They Felt the Video Was "Very Helpful" in Response to Second Question of Acceptability Questionnaire (Acceptability - Helpful)
Description: For the video intervention arm alone, we will administer 3-items assessing patients' comfort with watching the video, whether they find the video helpful in their understanding of the EOL care options, and whether they would recommend it to others. For the outcome of "helpful" we asked patients whether they felt the video was helpful by asking the question: "Was the video helpful in improving your understanding about your choices for medical care?". Response choices were on a Likert scale with answer choices as follows: 1) very helpful; 2) somewhat helpful; 3) a little helpful; 4) not helpful. We report below the percentage of patients who answered "very helpful".
Time Frame: Within 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Care Planning Video Decision Support Tool
Number analyzed (Participants) | 26
Participants | 19

7. Secondary Outcome: Number of Participants Who Answered That They Would "Definitely Recommend" the Video to Other Patients in Response to Third Question on Acceptability Questionnaire (Acceptability - Recommend to Others)
Description: For the video intervention arm alone, we will administer 3-items assessing patients' comfort with watching the video, whether they find the video helpful in their understanding of the EOL care options, and whether they would recommend it to others. For the outcome of "recommend to others" we asked patients whether they would recommend the video to other patients by asking the question: "Would you recommend the video to other patients with advanced liver disease who are facing a similar decision?". Response choices were on a Likert scale with answer choices as follows: 1) I would definitely recommend it; 2) I would probably recommend it; 3) I would probably not recommend it; 4) I would definitely not recommend it. We report below the percentage of patients who answered "I would definitely recommend it".
Time Frame: within 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Care Planning Video Decision Support Tool
Number analyzed (Participants) | 26
Participants | 24

ADVERSE EVENTS:
Time Frame: 12 months
Description: This study was a minimal risk study involving a video intervention tool. The only adverse event that was monitored for was serious distress by patients watching the video.
Arm/Group | Advanced Care Planning Video Decision Support Tool | Verbal Narrative Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT03557086/Prot_SAP_000.pdf